CLINICAL TRIAL: NCT06262919
Title: Observational Study to Assess Safety and Effectiveness of Dabrafenib and Trametinib in Patients With BRAF V600E Mutation-positive Unresectable Advanced or Recurrent Solid Tumor
Brief Title: Special Drug Use-results Surveillance of Tafinlar/Mekinist
Status: Recruiting | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CDRB436I1401
Record Dates: First submitted 2024-02-08; First posted 2024-02-16 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: BRAF V600E Mutation-positive Unresectable Advanced or Recurrent Solid Tumor
Keywords: Tafinlar; dabrafenib; Mekinist; trametinib; BRAF V600E mutation-positive unresectable advanced; solid tumor; Japan; recurrent
MeSH Terms: conditions — Recurrence | interventions — dabrafenib; trametinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Tafinlar/Mekinist: Patients with BRAF V600E mutation positive unresectable advanced or recurrent solid tumors treated with dabrafenib and trametinib as per Japanese Package Insert.
  Interventions: Drug: Tafinlar/Mekinist

INTERVENTIONS:
Drug: Tafinlar/Mekinist — There is no treatment allocation. Patients administered Tafinlar/Mekinist by prescription that have started before inclusion of the patient into the study will be enrolled.
  Other Names: Dabrafenib/trametinib

SUMMARY:
This is a prospective, multicenter, single-arm, non-interventional and observational J-PMS conducted by the central registration system and operated in Electronic data capture.

DETAILED DESCRIPTION:
In the Post-Marketing Surveillance (PMS), dabrafenib and trametinib are used as the marketed drugs. Registration of the corresponding patients is to be conducted by the central registered system under current medical practice.

Target number of adult patient is 65 (as the number of patients in the effectiveness analysis set).

Target number of pediatric patient is not determined. Estimated number of enrolled patients is approximately 20 (as the number of patients in the enrolled set)

The observation period for pediatric patients will last after the start of treatment until 8 years (planned, November 2031) after the approval of additional indications, regardless of discontinuation of the product, in order to collect long-term information from as many patients as possible during the reexamination period. The duration of observation for adult patients will be 1 year after the start of treatment with the product.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who have given written consent to cooperate in this surveillance
2. For patients aged < 18 years at the start of treatment with the product, their legally authorized representative must have given written informed consent for cooperation in this surveillance prior to patient enrollment.
3. Patients who start treatment with the product for BRAF-mutation-positive advanced/recurrent solid tumors (excluding colorectal cancer) after the approval of additional indications

Exclusion Criteria:

1. Patients who have received or are receiving a product containing the same ingredient as the product in any other study or research than this surveillance
2. Patients with BRAF-mutation-positive malignant melanoma
3. Patients with BRAF-mutation-positive non-small cell lung cancer
4. Patients with BRAF-mutation-positive hairy cell leukemia

Ages: 6 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients who used the product for the treatment of BRAF-mutation-positive advanced/recurrent solid tumors (excluding colorectal cancer) as per the package insert.
Sampling Method: Non-Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2024-02-09 (Actual); Primary Completion 2031-12-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
[Pediatric patients] Number of patients and incidence of adverse events/adverse reactions with respect to skeletal and sexual maturation | Up to 8 years
  To evaluate impairment in growth and development in pediatric patients (skeletal and sexual maturation) of dabrafenib and/or trametinib in pediatric patients under 18 years old in the post marketing phase.
[Adult patients] overall response rate (ORR) | 1 year
  The Overall Response Rate (ORR) is defined as the proportion of patients with a best OR of confirmed Complete Response (CR) or Partial Response (PR)

SECONDARY OUTCOMES:
[Pediatric patients] Incidence proportion of ORR | 1 year
  The Overall Response Rate (ORR) is defined as the proportion of patients with a best OR of confirmed Complete Response (CR) or Partial Response (PR)
[Pediatric and adult patients] Incidence proportion of PFS | 1 year
  Progression Free Survival (PFS) is the percentage of participants who did not have a progression event.
[Pediatric patients] Number of patients with changes in height and body weight and sexual maturation | Up to 8 years
  Number of pediatric patients with changes in height and body weight and sexual maturation is going to be collected

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (53):
- Japan (53):
  - Novartis Investigative Site, Nagakute, Aichi-ken
  - Novartis Investigative Site, Nagoya, Aichi-ken
  - Novartis Investigative Site, Toyohashi, Aichi-ken
  - Novartis Investigative Site, Toyota, Aichi-ken
  - Novartis Investigative Site, Daisen, Akita
  - Novartis Investigative Site, Chiba, Chiba
  - Novartis Investigative Site, Funabashi, Chiba
  - Novartis Investigative Site, Kashiwa, Chiba
  - Novartis Investigative Site, Fukuoka, Fukuoka
  - Novartis Investigative Site, Kurume, Fukuoka
  - Novartis Investigative Site, Fukuyama, Hiroshima
  - Novartis Investigative Site, Sapporo, Hokkaido
  - Novartis Investigative Site, Amagasaki, Hyōgo
  - Novartis Investigative Site, Kobe, Hyōgo
  - Novartis Investigative Site, Mito, Ibaraki
  - Novartis Investigative Site, Morioka, Iwate
  - Novartis Investigative Site, Kagoshima, Kagoshima-ken
  - Novartis Investigative Site, Sagamihara, Kanagawa
  - Novartis Investigative Site, Yokohama, Kanagawa
  - Novartis Investigative Site, Yokohama, Kanagawa-ku
  - Novartis Investigative Site, Kyoto, Kyoto
  - Novartis Investigative Site, Natori-shi, Miyagi
  - Novartis Investigative Site, Sendai, Miyagi
  - Novartis Investigative Site, Iida, Nagano
  - Novartis Investigative Site, Matsumoto, Nagano
  - Novartis Investigative Site, Yufu, Oita Prefecture
  - Novartis Investigative Site, Okayama, Okayama-ken
  - Novartis Investigative Site, Habikino, Osaka
  - Novartis Investigative Site, Izumisano, Osaka
  - Novartis Investigative Site, Osaka, Osaka
  - Novartis Investigative Site, Takatsuki, Osaka
  - Novartis Investigative Site, Kawagoe, Saitama
  - Novartis Investigative Site, Saitama, Saitama
  - Novartis Investigative Site, Sunto Gun, Shizuoka
  - Novartis Investigative Site, Shimotsuke, Tochigi
  - Novartis Investigative Site, Bunkyo Ku, Tokyo
  - Novartis Investigative Site, Bunkyo-ku, Tokyo
  - Novartis Investigative Site, Chuo Ku, Tokyo
  - Novartis Investigative Site, Minato-ku, Tokyo
  - Novartis Investigative Site, Setagaya-ku, Tokyo
  - Novartis Investigative Site, Shibuya City, Tokyo
  - Novartis Investigative Site, Shinjuku Ku, Tokyo
  - Novartis Investigative Site, Shinjuku-ku, Tokyo
  - Novartis Investigative Site, Wakayama, Wakayama
  - Novartis Investigative Site, Yamagata, Yamagata
  - Novartis Investigative Site, Akita
  - Novartis Investigative Site, Fukuoka
  - Novartis Investigative Site, Hiroshima
  - Novartis Investigative Site, Kochi
  - Novartis Investigative Site, Kyoto
  - Novartis Investigative Site, Okayama
  - Novartis Investigative Site, Osaka
  - Novartis Investigative Site, Shizuoka

IPD SHARING:
Plan to Share IPD: No